CLINICAL TRIAL: NCT01675349
Title: Biological Standardization of Chenopodium Album Allergen Extract to Determine the Biological Activity in Histamine Equivalent Prick (HEP) Units
Brief Title: Biological Standardization of Chenopodium Album Allergen Extract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Leti, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6062 -PR-PRI-195
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2012-08

CONDITIONS: Allergy to Chenopodium Album
Keywords: Standardization; Immunotherapy; Skin prick test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chenopodium album allergen extract (Experimental): Four concentrations of Chenopodium album allergen extract, together with a positive and negative control, using 10 mg/ml histamine dihydrochloride solution and a glycerinated phenol saline solution, respectively, will be tested in every patient in duplicate on the volar surface of the forearm. This test will be referred to as the Titrated Skin Prick test.
  Interventions: Biological: Prick test Chenopodium album allergen extract

INTERVENTIONS:
Biological: Prick test Chenopodium album allergen extract — This is an open, unblinded and non randomized biological as proposed by the Nordic Guidelines.
  Four concentrations of Chenopodium album allergen extract, together with a positive and negative control, using 10 mg/ml histamine dihydrochloride solution and a glycerinated phenol saline solution, respectively, will be tested in every patient in duplicate on the volar surface of the forearm. This test will be referred to as the Titrated Skin Prick test.
  Other Names: Chenopodium album allergen extract,

SUMMARY:
The objective of this study is to determine the biologic activity of a Chenopodium album allergen extract in histamine equivalent prick (HEP) units, in order to be used as in-house reference preparation (IHRP).

DETAILED DESCRIPTION:
This is an open, unblinded and non-randomized biological assay. The study design is a slight modification of the recommendations proposed by the Nordic Guidelines.

Four concentrations of Chenopodium album allergen extract, together with a positive and negative control, using 10 mg/ml histamine dihydrochloride solution and a glycerinated phenol saline solution, respectively, will be tested in every patient in duplicate on the volar surface of the forearm.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent, appropriately signed and dated by the subject (or legal representative, if applicable).
* Subject can be male or female of any race and ethnic group.
* Age > and =18 years and < and =60 years at the study inclusion day.
* Positive skin prick test with a standardized commercially available preparation of chenopodium album allergen extract.
* A positive test for specific IgE to chenopodium album (CAP-RAST major or equal to 2).
* Allergic symptoms during the pollen season of Chenopodium album.
* Medical history positive allergy inhalation (rhinitis and /or rhinoconjunctivitis and/or asthma) from Chenopodium album.

Exclusion Criteria:

* Immunotherapy in the past 5 years with an allergen preparation known to interfere with the allergen to be tested.
* Use of drugs that may interfere with the skin reactions (e.g., antihistamines).
* Treatment with any of the following medications: tricyclic or tetracyclic

  o IMAOs antidepressants,b-blockers or chronic use of corticosteroids or oral or use of corticoids both via oral or parenteral, in repeated patterns and intermittent (> 10 mg/día de prednisone or equivalent).
* Women who are pregnant or period of breastfeeding and women with a pregnancy test positive during the visit 2, prior to the prick test.
* Dermographism affecting the skin area at the test site at either study visit.
* Atopic dermatitis affecting the skin area at the test site at either study visit.
* Urticaria affecting the skin area at the test site at either study visit.
* Diseases of the immune system relevant clinically, both autoimmune and immunodeficiencies.
* Serious diseases not controlled that may increase the risk for the safety of the subjects involved in this study, including, but not limited to the following: heart failure, uncontrolled or severe respiratory diseases, endocrine diseases, clinically relevant kidney or liver diseases or hematological diseases.
* Participation in any other clinical trial within 30 days (or 5 times the biological half-life of the research of the study product, whichever is longer) prior to the inclusion of the subject in this clinical trial.
* Patients with diseases or conditions that limit the use of adrenaline (heart disease, severe hypertension, ..)
* Severe psychiatric, psychological or neurological disorders
* Abuse of alcohol, drugs or medicines in the previous year.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Wheal size area (mm2) on the skin at the site of the puncture during the immediate phase. | 15-20 min after application

CONTACTS AND LOCATIONS:
Overall Officials: Lena Erbiti, Study Chair — Laboratorios LETI, S.L.Unipersonal
Locations (2):
- Spain (2):
  - Hospital General de Elche, Alicante, Alicante
  - Centro Médico Adeslas, Córdoba, Córdoba